CLINICAL TRIAL: NCT05013034
Title: Fort Worth Clinical Sciences Working Group (FWCSWG) for COVID-19: Exploratory Regimen of Basiliximab for Treatment of Pulmonary Cytokine Storm in SARS-CoV-2 Hospitalized Adult Patients
Brief Title: Exploratory Regimen of Basiliximab for Treatment of Pulmonary Cytokine Storm in SARS-CoV-2 Hospitalized Adult Patients
Acronym: FWCSWG-IL-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fort Worth Clinical Sciences Working Group (Other)
Collaborators: TCU and UNTHSC School of Medicine (Other)
Responsible Party: Principal Investigator, Mohanakrishnan Sathyamoorthy MD, Chair, Fort Worth Clinical Sciences Working Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWCSWG-COVID19-01
Record Dates: First submitted 2021-08-18; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease; SARS-CoV2 Infection; Cytokine Storm
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome | interventions — Basiliximab

STUDY DESIGN:
Intervention Model Description: Number of Subjects A total of 300 subjects will be enrolled: 150 will be randomized to the basiliximab arm and 150 to the placebo arm in a 1:1 distribution.
  Treatment Assignments Qualified individuals will be randomized with a superiority design to either basiliximab (Simulect) or placebo. Study drug or placebo will be double blinded and administered on day 0 for all subjects. A second dose may be administered on Day 4 if first dose did not return the subject to a SpO2 ≥94% on room air.
  Criteria for Study Termination Although the FWCSWG intends to complete the study, the FWCSWG reserves the right to discontinue the study at any time for clinical or administrative reasons, or if required by regulatory agencies. If the FWCSWG discontinues the study, all study drugs will be discontinued and the investigator will be responsible for securing any alternative therapy to be administered, as appropriate.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Current Standard of Care) (Placebo Comparator): Current Standard of Care for SARS-CoV2 hypoxemic pulmonary diease
  Interventions: Drug: Placebo
- Basiliximab (Experimental): Basiliximab in addition to Current Standard of Care for SARS-CoV2 hypoxemic pulmonary diease
  Interventions: Drug: Basiliximab Injection

INTERVENTIONS:
Drug: Basiliximab Injection — Subjects will be given IV dosing with basiliximab up to a maximum of 2 treatments (day 0 and day 4) for all patients on study. Treatment for patients may stop for unacceptable side-effects, the Investigator's, or patient's decision to discontinue treatment or other reasons. Exclusion for second dose is first dose returned patient to SpO2 ≥94% on room air.
  Other Names: Simulect
  Arms: Basiliximab
Drug: Placebo — Subjects will be given IV dosing with placebo (1/2 normal saline) up to a maximum of 2 treatments (day 0 and day 4) for all patients on study. Treatment for patients may stop for unacceptable side-effects, the Investigator's, or patient's decision to discontinue treatment or other reasons. Exclusion for second dose is first dose returned patient to SpO2 ≥94% on room air.
  Arms: Placebo (Current Standard of Care)

SUMMARY:
To explore the efficacy of treatment of pulmonary cytokine storm induced by SARS-CoV2 with a monoclonal antibody to IL-2 (Basiliximab) in addition to current standard of care vs current standard of care with the primary efficacy endpoint being the proportion of subjects alive and free of ventilator support, defined as intubation and requiring mechanical ventilation, at Day 28 from time of randomization.

DETAILED DESCRIPTION:
The current pandemic driven by SARS-CoV2 creating the COVID-19 disease state is creating enormous healthcare challenges globally with limited treatment paradigms outside of supportive medical, and intensive care measures.

As the human population was entirely naïve to this viral pathogen, a particularly vigorous response of the immune cascade through cell-mediated mechanisms is a driving force behind the lethality of this disease in susceptible individuals. It is not presently understood why specific populations are at higher risk for disease state progression outside of traditional parameters such as age and pre-existing co-morbid health states. Furthermore, we lack a priori ways of identifying which SARS-COv2 infected patient may ultimately develop a "hyperactive" immune response that leads to the "cytokine storm" or "cytokine release syndrome", and the resultant cell, tissue, and organ system dysfunction.(1) Hypotheses in this area may include viral load phenomenon, aberration in immune/inflammatory regulatory check-points (JAK-STAT, JNK etc.), or underlying case dependent genetic factors (HLA etc.) influencing the immune system (2). Once the cytokine storm drives the clinical endpoint above, an affected patient who survives will become high risk for secondary pathogenic infection.

Intravenous remdesivir (3) along with dexamethasone (4, 5) have become standard of care therapeutics. The FDA recently provided emergency use authorization (EUA) for a novel SARS-COV2 neutralizing monoclonal antibody cocktail targeting the spike protein that docks with the ACE2 receptor on susceptible cells (Regeneron) (5). Rapid development of robust viral treatment strategies and vaccine development are the key strategies to managing SARS-COV2 in the long term. To this end, the FDA will be reviewing an EUA application for Pfizer's mRNA vaccine in early December, with similar review expected for Moderna's mRNA vaccine.

However, promising these developments are, thousands of patients are dying from cytokine storm mediated endpoints on a daily basis in the United States and across the world during the ongoing third wave/surge of COVID-19. There is broad recognition of this cytokine phenomenon, and in this era of targeted interleukin therapy for autoimmune disease states, a multitude of FDA approved monoclonal antibodies targeted to specific interleukins exist. Many institutions adopted IL-6 as a target for mitigation of the cytokine storm, and are utilizing tocilizumab (Actemra ®, Roche/Genentech) as a treatment (6) Sarilumab (Kevzara ®, Sanofi/Regeneron), another monoclonal Ab to IL-6, underwent rapid assessment for use in COVID-19(7). Both therapeutics did not meet primary specified endpoints in broader, Phase 2-3 studies.

These studies targeted the Th2/Tfh cytokine IL-6, as it plays a role in cytokine mediated inflammation in the lungs (9, 10) There is evidence that Il-6 can be induced within several hours by certain viral species (11) perhaps providing another reason why this was chosen as a target. Finally, this cytokine may serve as a target based on existing protocols to treat macrophage activation syndrome (MAS), and based on early evidence of cytokine expression patterns in patients infected with SARS-COV2 in Wuhan, PRC (2, 12-14). Classically, however, Th2/Tfh related cytokines are associated with antibody mediated immune memory and response, and though Th2/Tfh cytokines play a crucial role in acute inflammation, we have not seen protocols that target differentiating cytokines that drive Th0 to Th1 maturation, or Th1 specific cytokines. The Th1 cytokine profile is more consistently demonstrated in almost all early viral infection, and therefore, we view these cytokines as potential targets for therapy to prevent or mitigate the cytokine storm (Figure 1) (2, 12). Cytokine storm is a downstream manifestation of the viral induced host response that represents either failure of the initial host response to mitigate viral load, an uncontrolled late cytotoxic T-cell activity, or both. There is no evidence that targeted therapy against Th1 cytokines impairs the host response with strong clinical evidence supporting use in other EBV mediated secondary HLH syndromes (15).

The cytokine environment in which antigen primed T cells differentiate determines the subset that develops. In particular, IL-4 is essential for the development of Th2 response and IFN-gamma, IL-12 and IL-18 all are important in the development of Th1 cells. Th1 cells produce IL-2 and IFN-g, which in turn, promote the differentiation of fully cytotoxic T cells from CD8+ precursors.

A recent report published in Nature Medicine by Long et al. demonstrated a multi-fold higher expression of Th-1 cytokines, in particular, TNF alpha and IL-2, and significant expression of the IL-2 receptor subunit alpha in symptomatic COVID 19 patients in Wuhan.(16) A subsequent report published in Science Immunology by Lee et al. (17) demonstrated similar results through transcriptional and immuno-profiling techniques, and most recently a report in Nature (18) did the same. Therefore, among all immunomodulatory therapies, we view that targeting the Th1 response to be a key strategy. We propose targeting the IL-2R with Basiliximab.

Basiliximab (Simulect ®) is a monoclonal antibody against a subunit of IL-2 and is FDA approved for the treatment of acute renal transplant rejection, and is used off label in many other cases of transplant rejection mitigation.(2, 12) This agent has a long track record of safety and we believe among Th1 cytokine targets, to be a safe target for inhibition in SARS-COV2 induced cytokine storm.

Additional novel methodologies, including treatment with orally approved FDA approved JAK-STAT inhibitors (2) sirolimus (19-21) or calcineurin inhibitors (12) may serve as a broader opportunity to maintain suppression of inflammation following acute phase cytokine storm intervention with Basilixamab. One new area of interest is in complement mitigation, and inhibitors (eciluzimab) targeting this more teleologically more primal cascade may have a role (12, 22).

ELIGIBILITY:
Inclusion Criteria:

Subject Inclusion Criteria

1. Patient or legally authorized representative (LAR) willing and able to provide written or electronic or otherwise FDA-acceptable informed consent based on current FDA regulations.
2. Hospitalized male or non-pregnant female
3. RT-PCR confirmed SARS-CoV-2 using WHO consensus or validated primers
4. Meet the Following Criteria:

   1. Deficiency in Oxygenation as defined by the Berlin ARDS Criteria (27):

      Timing: Within 1 week of onset of symptoms Imaging: Bilateral pulmonary infiltrates

      Oxygenation (any):

      Mild: 200 mmHg < PaO2/FiO2 ≤ 300 mmHg Moderate: 100 mmHg < PaO2/FiO2 ≤ 200 mmHg Severe: PaO2/FiO2 ≤ 100 mmHg and
   2. Requiring oxygen support in the form of High Flow Nasal Cannula (HFNC), non-invasive positive pressure ventilation, intubation and mechanical ventilation, or initiation of ECMO and
   3. Any one or more of the following:

      1. Elevated CRP (>10 gm/dL)
      2. Elevated Ferritin (>1000)
      3. Neutrophil/lymphocyte ratio >3.3
5. Patient will receive current clinical standard of care. This includes inpatient use of remdesivir, dexamethasone, convalescent plasma, or pre-hospitalization outpatient treatment with casirivimab and imdevima
6. Age ≥ 18 years

Exclusion Criteria:

1. Off label use of other drugs
2. WOCBP unwilling to use acceptable birth control for 5 weeks, or male partner of a WOCBP unwilling to use male barrier method (condom) plus effective second method birth control for partner
3. Pregnant women
4. Pancytopenia

   1. Hgb< 8 g/dL (male) or < 7 g/dL (female)
   2. WBC<2.0 x 109/L
   3. PLT< 50 x 109/L

4) Enrollment in any study using immunomodulatory therapies (monoclonal antibodies, small molecule inhibitors etc. to interleukins or interleukin-receptor) 5) Any subjects who have received treatment with immunomodulators or immunosuppressant drugs, including but not limited to IL-6 inhibitors, TNF inhibitors, anti-IL-1 agents, and JAK inhibitors within 5 half-lives or 30 days (whichever is longer) prior to randomization.

6) Known/established systemic bacteremia (empiric antibiotics are allowed), uncontrolled viral infection besides the SARS-CoV-2 study disease, significant abscess in the opinion of the investigator, or any other finding that, in the opinion of the investigator, poses undue risk for treatment with basiliximab.

7) Any patient with multi-organ system failure or on intravenous vasopressor support 8) Do-not-resuscitate status at time of consent, or any contraindication to invasive mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | From time of randomization to Day 28
  1. Proportion of subjects alive and free of ventilator support, defined as intubation and requiring mechanical ventilation, at Day 28 from time of randomization

SECONDARY OUTCOMES:
Avoidance of escalation of O2 therapy | From time of randomization to Day 28
  Avoidance of escalation in oxygen therapy from the time of randomization to Day 28, defined as a binary endpoint, in which an increase from the baseline level of oxygen support to any of the following in the sequence listed below is considered an escalation, allowing for assessment of change in oxygen support at levels less than or greater than intubation and mechanical ventilation. Changes in level of oxygen therapy that occur prior to Day 28 are not accounted for in this endpoint.
  * Non-invasive positive pressure ventilation
  * Intubation and mechanical ventilation
  * Initiation of ECMO, with or without intubation and mechanical ventilation
  * Death
Overall Survival | From time of randomization to Day 28
  Overall survival, defined as proportion of subjects alive at Day 28 from time of randomization
ICU Free Survival | From time of randomization to Day 28
  ICU-free survival, defined as proportion of subjects alive and not requiring ICU hospitalization at Day 28 from time of randomization
ECMO Free Survival | From time of randomization to Day 28
  ECMO-free survival, defined as proportion of subjects alive and not requiring ECMO support at Day 28 from time of randomization
Overall Survival at 90 days | From time of randomization to Day 90
  Overall survival, defined by time to event analysis at Day 90
Ventilator-free survival at 90 days | From time of randomization to Day 90
  Ventilator-free survival, defined by time to event analysis at Day 90

OTHER OUTCOMES:
ICU length of stay | From time of randomization to Day 90
  Exploratory
Hospital length of stay | From time of randomization to Day 90
  Exploratory
ICU length of stay + death composite endpoint | From time of randomization to Day 90
  Exploratory
Hospital length of stay + death composite endpoint | From time of randomization to Day 90
  Exploratory
Improvement in 8-point ordinal scale | From time of randomization to Day 28
  Improvement in 8-point ordinal scale
Decline in serum albumin | From time of randomization to Day 28
  Decline in serum albumin
proportion alive and free of ventilator support stratified by IV dexamethasone | From time of randomization to Day 28
  proportion alive and free of ventilator support stratified by IV dexamethasone

CONTACTS AND LOCATIONS:
Overall Officials: mohanakrishnan sathyamoorthy, Principal Investigator — FWCSWG

IPD SHARING:
Plan to Share IPD: Undecided